CLINICAL TRIAL: NCT03635853
Title: Identification of Compound Isolated From Cock's Comb and Its Effect on Arsenical Palmar Keratosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Hazera Sharmin, Resident, Dept. of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No. BSMMU/2018/2966
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Improvement of Keratotic Nodular Size

STUDY DESIGN:
Intervention Model Description: a single group of patients with palmar arsenical keratosis are given the drug, under study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with palmar arsenical keratosis (Experimental): patients are given an ointment containing extract from cock's comb twice daily for three months
  Interventions: Drug: drug containing extract from cock's comb

INTERVENTIONS:
Drug: drug containing extract from cock's comb — a container containing 25 mg of ointment having extract from cock's comb as active ingredient two times daily for 3 months

SUMMARY:
Arsenicosis is a massive public health hazard in Bangladesh. Prolonged consumption of water containing high concentration arsenic leads to arsenicosis which is characterized by dermatological features i.e. diffuse melanosis , spotted melanosis and keratosis. Cock's comb is rich in hyaluronic acid, chondroitin sulfate A, B, C and heparin. Hyaluronic acid is a hydrophilic molecules and is a constituent of wound extracellular matrix and facilitate wound healing.This work is aimed to identify the component that is effective in palmar arsenical keratosis.

DETAILED DESCRIPTION:
Groundwater contamination caused by inorganic arsenic is a massive public health hazard in Bangladesh. Prolonged consumption of water containing high concentration arsenic leads to chronic arsenic poisoning which is characterized by dermatological features i.e. diffuse melanosis followed by spotted melanosis hyperpigmentation and keratosis.

Until now there is no internationally accepted treatment for arsenical keratosis. Some authors suggest long-term administration of vitamin and mineral and topical application of salicylic acid, propylene glycol and neem may be effective. Cock's comb extract contains hyaluronic acid, chondroitin sulfates A, B and C, heparin, hexosamine and water. Study with cock's comb extract in the treatment of arsenical keratosis was done in the Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University and was found effective. Therefore, the purpose of this study will be identification of compound isolated from cock's comb and its effect on palmar arsenical keratosis. After obtaining Institutional review board clearance, on the basis of inclusion and exclusion criteria, 40 patients with moderate to severe palmar arsenical keratosis will be enrolled from arsenic affected area located at Kamalla Union of Muradnagar Upazilla, Comilla. The study will be open phase II clinical trial. After enrollment, patients will be informed about the purpose as well as harmful and beneficial effects of the study. Informed written consent, detail history, clinical examination, photographs of the palm and water and nail samples will be collected before starting recruitment to confirm arsenicosis. For identification of compound present in the cock's comb thin layer chromatography and nuclear magnetic resonance will be done. Cytotoxic effects of the cock's comb extract will be analyzed by using brine shrimp assay. Cream will be prepared from cock's comb extract and supplied to the patient at an interval of 2 weeks to apply on palmar keratotic nodule with clean fingertip by rubbing gently at night for 12 weeks. Adherence of the cream and side effects will be monitored routinely through phone and during visit at field level. Improvement will be assessed by measuring the palmar keratotic nodular size with the help of slide calipers. The mean score of the nodular size before and after treatment will be done. Statistical analysis will be conducted by paired t test. The result will be presented in tabulated forms and bar diagrams.

ELIGIBILITY:
Inclusion Criteria:

* drinking arsenic contaminated water (>50 microgram/litre) for more than 6 months patients with moderate to severe arsenical palmar keratosis patients voluntarily agreed to participate patient did not receive topical application of any drug for the last three months

Exclusion Criteria:

* patient who received any treatment of arsenicosis within last three months patient with diagnosed skin disease, like-atopic dermatitis and psoriasis any diagnosed systemic diseases, inflammatory disease and infectious condition that affect the skin, for example- diabetes mellitus, SLE and hepatitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-16 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
changes in keratotic nodular size | three months
  palmar arsenical keratosis will be measured before and after applying interventions

CONTACTS AND LOCATIONS:
Overall Officials: Hazera Sharmin, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Kamalla, community clinic, Comilla, Muradnagar, Bangladesh